CLINICAL TRIAL: NCT02997267
Title: The Early Closure of the Protective Ileostomy After Low Anterior Resection Enables Correct Start of Chemotherapy
Brief Title: Early Closure of Protective Ileostomy in Rectal Cancer Patients
Acronym: ECPIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanley Dudrick's Memorial Hospital (Other)
Responsible Party: Principal Investigator, Stanislaw Klek, Head of the Department, Stanley Dudrick's Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zespolenia
Record Dates: First submitted 2016-12-05; First posted 2016-12-20 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early closure (Experimental): Closure of the ileostomy 14 days after the primary operation, in which it was created.
  Interventions: Procedure: Closure of the ileostomy
- Late closure (Active Comparator): Closure of the ileostomy more than 90 days after the primary operation, in which it was created.
  Interventions: Procedure: Closure of the ileostomy

INTERVENTIONS:
Procedure: Closure of the ileostomy — Surgical closure of the protective ileostomy (reconnection of intestinal loops)

SUMMARY:
The aim of the study was to compare the restoration of the GI tract by the closure of protective ileostomy after low anterior resection for rectal cancer after 14 days and more than 3 months.

DETAILED DESCRIPTION:
The closure of the protective ileostomy created during the low anterior resection for rectal cancer to protect the colo-rectal anastomosis is inevitable to restore the continuity of the gastrointestinal tract. It usually takes place several months after the primary surgery, because the patients starts chemotherapy and cannot undergo the procedure during the therapy. It results in the relative low quality of life of the patient, as well as often leads to complications. Therefore, it seem reasonable to close the stoma as soon as possible to take the burden off patient.

It is well known that the healing process of the anastomosis runs in the three phases, but only two first are crucial for the clinical result. The second takes place between 5th and 14th postoperative day. Therefore it should be possible to perform successful restoration of the GI tract already after two weeks after operation, and not after many moths.

The aim of the study was to compare the restoration of the GI tract after 14 days and more than 3 months, so to compare the traditional and early strategy.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 year old
* the presence of the protective ileostomy created during the low anterior resection to protect the colo-rectal anastomosis

Exclusion Criteria:

* the presence of the protective ileostomy created during any other procedure than the low anterior resection to protect the colo-rectal anastomosis
* age < 18 yo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Number of postoperative fistulas | 3 months after surgery
  number of patients with the fistula of the anastomosis

SECONDARY OUTCOMES:
Timing of anticancer therapy | 3 months after surgery
  Time to the beginning of adiuvant chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Stanley Dudrick's Memorial Hospital, Skawina, Poland

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.